CLINICAL TRIAL: NCT00747357
Title: The Paclitaxel-Eluting PTCA-Balloon Catheter in Combination With a Cobalt-Chromium Stent to Treat Coronary Artery Disease in a Real World Scenario
Brief Title: INDICOR The Paclitaxel-Eluting PTCA-Balloon Catheter in Combination With a Cobalt-Chromium Stent
Acronym: INDICOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ralf Degenhardt, PhD (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor-Investigator, Ralf Degenhardt, PhD, Data Manager, Heart Centre Rotenburg
Organization: Heart Centre Rotenburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBM-VS-57INDICOR/CRI/07-02/n-c
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Heart Diseases
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Balloon first
  Interventions: Device: Drug Eluting Balloon SeQuent Please
- 2 (Experimental): Stent First
  Interventions: Device: Drug Eluting Balloon SeQuent Please

INTERVENTIONS:
Device: Drug Eluting Balloon SeQuent Please — Drug Eluting Balloon is followed by Bare Metal Stent
  Other Names: SeQuent® Please DEB
  Arms: 1
Device: Drug Eluting Balloon SeQuent Please — Bare Metal Stent followed by Drug Eluting Balloon
  Other Names: SeQuent® Please DEB
  Arms: 2

SUMMARY:
The INDICOR study is a controlled, prospective, multicenter, randomized, two arm phase-II real world study assessing the acute, 6 months, and 12 months and 3 year outcome of cobalt-chromium stent (Coroflex Blue) deployment followed by Paclitaxel-eluting PTCA-balloon dilatation (SeQuent Please) and of Paclitaxel-eluting PTCA-balloon dilatation (SeQuent Please) followed by cobalt-chromium stent (Coroflex Blue) deployment for the treatment of de-novo and restenotic lesions in native coronary arteries. The study will be conducted in India.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the efficacy and safety of cobalt-chromium stent (Coroflex Blue) deployment followed by Paclitaxel-eluting PTCA-balloon dilatation (SeQuent Please) and of Paclitaxel-eluting PTCA-balloon dilatation (SeQuent Please) followed by cobalt-chromium stent (Coroflex Blue) deployment in a real world scenario including up to two de-novo or restenotic lesions ( no in-stent restenoses) in two different native coronary arteries (reference diameter: 2.5mm and 4.0mm, length of stenosis 10mm and 25mm) for procedural success and preservation of vessel patency up to 3 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina pectoris (CCS class 1-3) or with unstable angina pectoris (Braunwald class 1-2, A-C) or documented ischemia or with documented silent ischemia
* Patients eligible for coronary revascularization by means of PCI
* Patients suitable for coronary revascularization of any sort (balloon angioplasty, device-assisted balloon-angioplasty or coronary artery bypass grafting)
* Patients must be older then 18 years of age
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 6 months follow-up.
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 6 months angiographic follow-up
* Patients must agree to undergo the 1 year and 3 year clinical follow-up

Lesion Related (relates to up to 2 stenoses in two different coronary arteries to be treated per protocol)

* Reference diameters ranging from 2.5 mm to 4.0 mm and length of stenosis from 10 mm to ≤ 25 mm
* Diameter stenosis pre procedure must be either more then 70 % or more then 50 % if ischemia corresponding to the target lesion is documented either by exercise stress ECG, stress echocardiography, or scintigraphy
* Coverage of the target lesion must be intended and possible by a single Paclitaxel-eluting balloon

Exclusion Criteria:

Patient Related

* Patients with acute (< 24 h) or recent (≤ 48 hours) myocardial infarction
* Patients with unstable angina pectoris (Braunwald class 3)
* Patients with severe congestive heart failure
* Patients with severe heart failure NYHA IV
* Patients demonstrating clinical signs of cardiogenic shock at the time of the procedure (systolic blood pressure of less than 80 mm Hg requiring inotropic support, IABP and/or fluid challenge).
* Patients with severe valvular heart disease
* Women who are pregnant or lactating
* Patients with life expectancy of less than five years or factors making clinical follow-up difficult
* Patients with bleeding diathesis in whom anticoagulation or anti-platelet medication is contraindicated
* Patients who had a cerebral stroke < 6 months prior to the procedure
* Patient participates in other clinical trials involving any investigational device or drug
* Untreated hyperthyroidism
* Patient has presence or history of severe renal failure (GFR<30ml/min) and is therefore not eligible for angiography. Patient's serum creatinine levels must be documented
* Post transplantation of any organ or immune suppressive medication
* Other disease to jeopardize follow-up (e.g., malignancy)
* Addiction to any drug or to alcohol
* Patients with any type of surgery during the week preceding the interventional procedure
* Patients with percutaneous coronary intervention during the six months prior to enrollment into this study

Lesion Related

* Evidence of extensive thrombosis within target vessel before the intervention
* Side branch > 2 mm in diameter originating from the lesion
* Percutaneous coronary intervention of venous graft
* Target segment is occluded of (i.e., acute or chronic)
* In-stent restenosis (restenoses in non-stented segments are permitted)
* Ostial lesion within 2 mm of vessel origin
* Patients with another coronary stent implanted previously into the target vessel proximal to the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Late lumen loss at 6 months in-segment and in-stent for each treated coronary stenosis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Upendra kAUL, Dr., Principal Investigator — Fortis Flt.Lt.Rajan Dhall Hospital, New Delhi, India
Locations (1):
- Upendra Kaul, New Delhi, India